CLINICAL TRIAL: NCT04132323
Title: Clinical Efficacy of Low Concentrate Detergents Versus Hypertonic Glucose for the Treatment of Telangiectasia: a Prospective Randomized Clinical Trial
Brief Title: Low Concentrate Detergents Versus Hypertonic Glucose for the Treatment of Telangiectasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derzhavin Tambov State University (Other)
Responsible Party: Principal Investigator, Oksana Bukina, Director, Clinical Research, Derzhavin Tambov State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A001203
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-03

CONDITIONS: Sclerotherapy
Keywords: sclerotherapy, hypertonic glucose, sodium tetradecyl sulfate
MeSH Terms: interventions — Sclerotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- hypertonic glucose (Active Comparator): * to take photo of problem area in the patient's standing position in the room with artificial lighting using the iPhone 6s and above, Samsung Galaxy S7 and above from a distance of 20 cm.
  * to measure the maximum diameter of telangiectasia using the Dermatoscope scale.
  * to inject the 75% glucose, with a 2 ml luer-lock syringe through 30 G needle in telangiectasia until the vessel disappears.
  Interventions: Procedure: Sclerotherapy
- 0.05% sodium tetradecyl sulfate (Active Comparator): * to take photo of problem area in the patient's standing position in the room with artificial lighting using the iPhone 6s and above, Samsung Galaxy S7 and above from a distance of 20 cm.
  * to measure the maximum diameter of telangiectasia using the Dermatoscope scale.
  * to inject the 0.05% sodium tetradecyl sulfate with a 2 ml luer-lock syringe through 30 G needle in telangiectasia until the vessel disappears.
  Interventions: Procedure: Sclerotherapy
- 0.1% sodium tetradecyl sulfate (Active Comparator): * to take photo of problem area in the patient's standing position in the room with artificial lighting using the iPhone 6s and above, Samsung Galaxy S7 and above from a distance of 20 cm.
  * to measure the maximum diameter of telangiectasia using the Dermatoscope scale.
  * to inject the 0.1% sodium tetradecyl sulfate with a 2 ml luer-lock syringe through 30 G needle in telangiectasia until the vessel disappears.
  Interventions: Procedure: Sclerotherapy
- 0.15% sodium tetradecyl sulfate (Active Comparator): * to take photo of problem area in the patient's standing position in the room with artificial lighting using the iPhone 6s and above, Samsung Galaxy S7 and above from a distance of 20 cm.
  * to measure the maximum diameter of telangiectasia using the Dermatoscope scale.
  * to inject the 0.15% sodium tetradecyl sulfate with a 2 ml luer-lock syringe through 30 G needle in telangiectasia until the vessel disappears.
  Interventions: Procedure: Sclerotherapy

INTERVENTIONS:
Procedure: Sclerotherapy — Examination, photographing, inclusion in the study, signing of informed consent, randomization, diameter measurement, sclerotherapy according to the randomization group

SUMMARY:
Using of low concentrate sodium tetradecyl sulfate for sclerotherapy of telangiectasias should be no less effective than hypertonic glucose, and have a comparable frequency of adverse events.

DETAILED DESCRIPTION:
For sclerotherapy of telangiectasias are used detergents. These are aggressive substances, which have a high frequency of adverse events. According to histological studies the safest concentration for the treatment of telangiectasias is less than that specified in the official instructions. The concentration of sodium tetradecyl sulfate 0.15% was effective and did not cause any adverse reactions in the treatment of telangiectasias from 0.8 to 1 mm in diameter. Small telangiectases (0.5 mm or less) require the treatment with the less aggressive sclerosing agent. Perhaps, the sodium tetradecyl sulfate 0.15%, 0.1% or even 0.05% and hypertonic glucose may be more effective and safe in this situation.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* single primary or secondary telangiectasias unrelated to the reticular veins
* signed informed consent to participate in the study

Exclusion Criteria:

* telangiectasias associated with reticular veins
* diabetes mellitus
* pregnancy or lactation
* malignant neoplasms
* inability or unwillingness of the patient to wear compression stockings
* hypersensitivity to one of the drugs
* concomitant diseases: bronchial asthma, severe liver and kidney disease, acute thrombosis and thrombophlebitis, infection of the skin and/or soft tissues, infectious diseases, arteriosclerosis, diabetic angiopathy, heart defects requiring surgery, fever, toxic hyperthyroidism, obesity, tuberculosis, sepsis, violation of the cellular composition of the blood, all diseases requiring bed rest, heart disease with decompensation phenomena, known hereditary thrombophilia.
* period after treatment of alcoholism
* reception of oral contraceptives
* sedentary lifestyle

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Disappearance of the telangiectasia | 2 months
  The clearing of the vessels on the six-point scale (from 0 to 5 points): 5 - total disappearance of the matting (100% efficacy), 4 - disappearance of around 80%, 3 - disappearance of around 60%, 2 - disappearance of around 40%, 1 - disappearance of around 20%, 0 - no changes.

SECONDARY OUTCOMES:
Pain during the procedure: visual analog scale | immediately after the procedure
  Estimate of the pain on visual analog scale. Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal 10 cm length: "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).
Patient Satisfaction After Treatment | 2 months
  Assessment of patient satisfaction on the 3-point scale :
  * no result (0 points),
  * incomplete satisfaction (1 point),
  * complete satisfaction (2 points)

CONTACTS AND LOCATIONS:
Overall Officials: Oksana Bukina, PhD, Principal Investigator — Derzhavin Tambov State University
Locations (1):
- Bukina Oksana Vasilyevna, Tambov, Russia

IPD SHARING:
Plan to Share IPD: Yes
The study data are available to all investigators in the chronic vein disease registry.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 25 October 2019 to 25 December 2021
URL: https://www.venousregistry.org/index.php?u=1

REFERENCES:
- [Result] Bush R, Bush P. Evaluation of sodium tetradecyl sulfate and polidocanol as sclerosants for leg telangiectasia based on histological evaluation with clinical correlation. Phlebology. 2017 Aug;32(7):496-500. doi: 10.1177/0268355516673768. Epub 2016 Oct 12. PMID 27738241
- [Result] Rabe E, Schliephake D, Otto J, Breu FX, Pannier F. Sclerotherapy of telangiectases and reticular veins: a double-blind, randomized, comparative clinical trial of polidocanol, sodium tetradecyl sulphate and isotonic saline (EASI study). Phlebology. 2010 Jun;25(3):124-31. doi: 10.1258/phleb.2009.009043. PMID 20483861
- [Result] Parlar B, Blazek C, Cazzaniga S, Naldi L, Kloetgen HW, Borradori L, Buettiker U. Treatment of lower extremity telangiectasias in women by foam sclerotherapy vs. Nd:YAG laser: a prospective, comparative, randomized, open-label trial. J Eur Acad Dermatol Venereol. 2015 Mar;29(3):549-54. doi: 10.1111/jdv.12627. Epub 2014 Jul 28. PMID 25069999
- [Result] Munia MA, Wolosker N, Munia CG, Chao WS, Puech-Leao P. Comparison of laser versus sclerotherapy in the treatment of lower extremity telangiectases: a prospective study. Dermatol Surg. 2012 Apr;38(4):635-9. doi: 10.1111/j.1524-4725.2011.02226.x. Epub 2011 Dec 30. PMID 22221551
- [Derived] Bukina OV, Sinitsyn AA, Efremova OI, Pelevin AV. Low concentration of sodium tetradecyl sulfate and hypertonic glucose solution for the treatment of telangiectasia: A prospective randomized clinical trial. Phlebology. 2023 Oct;38(9):622-627. doi: 10.1177/02683555231191969. Epub 2023 Jul 30. PMID 37519033
- Available data/document: Study Protocol — https://www.venousregistry.org/index.php?f=1&id=97